CLINICAL TRIAL: NCT07254169
Title: The Efficacy and Safety of Herbal Medicine Treatment Strategy for Patients With Post-Accident Fatigue: A Pragmatic Randomized Controlled Pilot Clinical Trial
Brief Title: The Efficacy and Safety of Herbal Medicine Treatment Strategy for Patients With Post-Accident Fatigue
Acronym: TA fatigue
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-CT-2025-12; Jaseng Medical Foundation (Other: Jaseng Medical Foundation)
Record Dates: First submitted 2025-11-20; First posted 2025-11-28 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Post-traffic Accident Fatigue
Keywords: Fatigue Herbal medicine
MeSH Terms: interventions — Phytotherapy; Educational Status

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education plus herbal medicine group (Experimental): An informational booklet will be distributed and a brief training session will be provided at the time of study registration.
  The informational booklet will focus on providing information, including the definition and causes of fatigue, post-traumatic fatigue, and the impact of dietary habits and alcohol on fatigue.
  If necessary, acupuncture, moxibustion, herbal acupuncture, and Chuna therapy can be provided for post-traumatic treatment of other aftereffects besides fatigue.
  Interventions: Procedure: Herbal medicine; Procedure: Education
- Education-only group (Active Comparator): At the time of study registration, informational pamphlets will be distributed and brief training will be provided.
  If necessary, acupuncture, cupping therapy, herbal acupuncture, and Chuna therapy can be provided to treat aftereffects other than fatigue after a traffic accident.
  The clinician will prescribe a 14-day supply of herbal medicine based on the patient's diagnosis. Subjects in the herbal medicine group will take the herbal medicine orally twice daily for a total of 28 days during the treatment period.
  This study is a practical clinical trial and has no restrictions on the type of herbal medicine used. Prescriptions are made at the discretion of the medical staff, with the primary goal of alleviating fatigue. All prescriptions are written by a Korean medicine doctor with at least five years of clinical experience. After the prescriptions are issued, the herbal medicines are delivered to the participants via courier and consumed. Participants are instructed to store all herba
  Interventions: Procedure: Education

INTERVENTIONS:
Procedure: Herbal medicine — Herbal medicine treatment is a treatment using complex extract of medicinal herbs prescribed by a Korean medicine doctor who has completed specialized education to diagnose the health condition and symptoms of patients
  Arms: Education plus herbal medicine group
Procedure: Education — Educational materials will be distributed and training will be provided on managing daily life to alleviate fatigue. The information-based program will cover topics such as the definition and causes of fatigue, post-traumatic fatigue, and the impact of dietary habits and alcohol on fatigue.

SUMMARY:
This study is a pragmatic randomized controlled pilot clinical trial aimed at evaluating the efficacy and safety of herbal medicine treatment strategy for patients with post-traffic accident fatigue, using an education-only group as the control.

DETAILED DESCRIPTION:
0. Background Over three million traffic accidents occur annually across OECD countries, often resulting in fatigue, insomnia, and dizziness that persist beyond the acute phase. Post-accident fatigue is common even after mild injuries and can greatly hinder recovery and daily functioning. In Korean traditional medicine, it is viewed as a deficiency of qi and blood, for which herbal medicine treatment is used to restore vitality. This study aims to assess whether combining herbal medicine with education improves post-accident fatigue and to explore related body composition changes.

1. Patient Recruitment and Screening Phase

1. Patient Recruitment Forty patients meeting the inclusion/exclusion criteria will be recruited starting from the date of IRB registration. Researchers will use block randomization to allocate participants. After obtaining written consent from patients who meet the criteria, they will be assigned to the study. The probability of assignment to each group will be 1:1.
2. Allocation Concealment and Blinding Since blinding is not feasible for this study, it will be conducted as an open-label clinical trial. However, assessor blinding will be implemented. The evaluator, who will not participate in the intervention and will be blinded to group allocation, will conduct assessments in a separate space before the intervention. This role will be performed by a research nurse or a specialist in training.

2. Treatment and Evaluation Phase

1. Control and Experimental Groups

   - The test group will be divided into the "medicinal herbal medicine group," and the control group will be the "education-only group."

   - To study the additional effects of herbal medicine treatment while maintaining the same conditions for both groups, both groups will receive educational brochures as follows:
   * Subjects in both groups will receive an informational brochure and brief training at their first visit. The brochure will provide information-focused explanations, including the definition and causes of fatigue, post-traumatic fatigue, and the impact of dietary habits and alcohol on fatigue.
   * Subjects in both groups will be eligible to receive acupuncture, cupping therapy, pharmacopuncture, and Chuna therapy, if necessary, to treat aftereffects other than fatigue after a traffic accident. The type and method of treatment will be selected within the scope of current clinical practice at the relevant research institution, based on the subject's symptoms and the clinician's judgment. However, herbal medicine treatment aimed at alleviating traffic accident aftereffects will not be permitted during the study period due to concerns about potential confusion with the interventions in this study. - The supplement group will receive additional supplements based on the medical team's diagnosis and take them twice daily for a total of 28 days.
2. Study Duration and Observation Points

   - The study period for the subjects will be 12 weeks, including a 4-week treatment period and an 8-week follow-up period.
   * The baseline will be the study enrollment date (Week 0), and the primary endpoint will be Week 5.
   * Data will be collected during the treatment period (Weeks 1 and 3), and the follow-up visits (Weeks 5 (primary endpoint), 8, and 12).
3. Data Collection for Evaluation i. Primary Outcome

   - (1) FSS-K (Fatigue Severity Scale - Korean version)

   - The primary outcome is the FSS-K at Week 5, the end of the treatment intervention.

   - The assessment will be conducted at screening, enrollment, and assignment, Weeks 1 and 3 of the treatment period, and at follow-up visits at Weeks 5, 8, and 12.

   ii. Secondary Outcome

   - The following indicators will be assessed at visits during the treatment period (Weeks 1 and 3) and at follow-up visits (Weeks 5 (primary endpoint), 8, and 12).

   - (1) CFQ-K (Chalder Fatigue Questionnaire - Korean version)

   - (2) ISI-K (Insomnia Severity Index - Korean version)

   - (3) K-BDI (Beck Depression Inventory - Korean version)

   - (4) Quality of Life Assessment Scale (EQ-5D-5L)

   - (5) Body Fat Percentage
   * (6) Skeletal Muscle Mass
   * (7) Phase Angle
   * (8) Extracellular Water Ratio
   * (9) Adherence
   * (10) Adverse Effects

     3. Follow-Up Phase After the 4-week treatment period, the subjects will be followed up for 8 weeks to assess symptom changes. Both groups will undergo follow-up visits at 5, 8, and 12 weeks from the date of enrollment, assessing the primary outcome (FSS-K), secondary outcomes (CFQ-K, ISI-K, K-BDI, EQ-5D-5L, body fat percentage, skeletal muscle mass, phase angle, extracellular water content, and medication compliance), and adverse events, identical to those observed during the treatment period.

   The follow-up period after 5 weeks will have a time window of ±5 days. The follow-up period after 8 and 12 weeks will have a time window of ±7 days.

   Both groups will undergo blood tests at 5 weeks from the date of enrollment. The blood test items will be identical to those used during the screening period.

4. Monitoring The principal investigator or a co-investigator with medical judgment, authorized by the principal investigator, will maintain the integrity of the research data and collect and review safety data for the study subjects. Monitoring will be conducted every six months.

1. The safety and rights of the subjects are reported.
2. The clinical study is conducted in compliance with the currently approved research protocol and research management standards.
3. The data are reliable, accurate, and safe.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 40 to 69 years.
* Patients who have been in a traffic accident for 12 to 24 weeks.
* Patients with an average score of 4 or higher on the FSS-K questionnaire.
* Participants who voluntarily agreed to participate in the study and signed a consent form.

Exclusion Criteria:

* Participants diagnosed with and receiving treatment for a specific disease that may cause fatigue (cancer, anemia, thyroid dysfunction, etc.).
* Participants with clinically significant abnormalities in blood tests that may be a major cause of fatigue.
* Participants taking herbal medicine for fatigue relief or have taken health supplements for fatigue relief within the past two weeks.
* Participants with other chronic conditions that may interfere with the treatment effect or interpretation of results: stroke, myocardial infarction, kidney disease, active hepatitis, diabetic neuropathy, dementia, epilepsy, etc.
* Participants currently taking steroids, immunosuppressants, psychiatric medications, or other medications that may affect the study results.
* Participants who are not suitable for herbal medicine treatment. Unsafe: Patients with conditions that may affect drug intake or absorption, those with digestive problems following surgery related to such conditions, or those with severe liver or kidney disease (AST, ALT, γ-GTP, and serum creatinine levels greater than twice the upper limit of normal during screening).
* Are pregnant, planning to become pregnant, breastfeeding, or may be pregnant (e.g., recent missed menstrual periods, irregular menstrual cycles, not using contraception, recently had sexual intercourse, or the investigator determines through medical history that pregnancy is possible).
* Participating in research studies other than observational studies without therapeutic intervention.
* Difficulty completing the consent form.
* Other circumstances in which participation in a clinical trial is deemed difficult by the investigator.

Ages: 40 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
FSS-K (Fatigue Severity Scale - Korean version) | Screening, Week 1, Week 3, Week 5, Week 8, Week 12
  The FSS-K assesses fatigue levels over the past week on a scale of 1 to 7, with nine questions. The final FSS score is calculated by adding the scores for each item and dividing by 9, resulting in an average. Higher scores indicate greater fatigue.

SECONDARY OUTCOMES:
CFQ-K (Chalder Fatigue Questionnaire - Korean version) | Week 1, Week 3, Week 5, Week 8, Week 12
  The CFQ-K is a 14-item self-report scale divided into two domains: physical fatigue symptoms (8 items) and mental fatigue symptoms (6 items). Each item has five response options ('none', 'better than usual', 'as usual', 'worse than usual', 'very bad') and is scored from 0 to 4. Each subscale score is calculated by summing the scores of all items in that domain, and the overall fatigue score is calculated by summing the scores of all 14 items, with higher scores indicating more severe fatigue.
ISI-K (Insomnia Severity Index - Korean version) | Week 1, Week 3, Week 5, Week 8, Week 12
  ISI-K is a questionnaire that evaluates the severity of insomnia and consists of 5 questions, each of which is scored from 0 (no insomnia) to 4 (most severe insomnia).
K-BDI (Beck Depression Inventory - Korean version) | Week 1, Week 3, Week 5, Week 8, Week 12
  The K-BDI consists of 21 items covering the cognitive, emotional, motivational, and physical symptom domains of depressive symptoms. Each item consists of four options describing the severity of depressive symptoms. Scores range from 0 (1) to 3 (4), and each item's score is summed to obtain a total score. Scores range from 0 to 63.
5-Level EuroQol-5 Dimension (EQ-5D-5L) | Week 1, Week 3, Week 5, Week 8, Week 12
  The 5-Level EuroQol-5 Dimension (EQ-5D-5L) is one of the most widely used indirect measurement methods for calculating the quality weight of a specific health state. It evaluates health status from multiple perspectives and utilizes pre-assigned preference scores for each functional level to indirectly calculate the quality weight of a particular health condition. The EQ-5D-5L consists of five items, each addressing the degree of mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item is assigned a specific weight based on its level, and a preference score calculation formula is provided using these weights and constants.
Body Fat Percentage | Week 1, Week 3, Week 5, Week 8, Week 12
  This refers to the percentage of body fat relative to body weight. Obesity is more appropriately assessed by the percentage of body fat relative to body weight than by the actual body fat mass. For men, the standard body fat percentage is 15% of standard body weight, and for women, it is 23% of standard body weight.
Skeletal muscle mass | Week 1, Week 3, Week 5, Week 8, Week 12
  This is the amount of muscle attached to the skeleton, excluding involuntary muscles such as visceral muscles.
Phase Angle | Week 1, Week 3, Week 5, Week 8, Week 12
  This represents the resistance across the cell membrane, expressed as an angle. The higher the structural stability of the cell, the higher the value. A healthy cell exhibits a high value, while a deteriorating cell membrane condition results in a value closer to 0.
Extracellular Water Ratio | Week 1, Week 3, Week 5, Week 8, Week 12
  This represents the ratio of intracellular water (ICW) to extracellular water (ECW), indicating body water balance. The standard range is 0.36 to 0.39.
Adherence | Week 5
  To assess treatment compliance, for participants in the herbal medicine treatment group, the cumulative number of herbal medicine packs prescribed and the number of unused herbal medicine packs are recorded in the CRF for those receiving supplements at Week 5.
Adverse Event (AE) | Week 3, Week 5, Week 8, Week 12
  An adverse event refers to any undesirable and unintended objective sign, subjective symptom, or disease that occurs after a clinical trial procedure, and it does not necessarily have to have a causal relationship with the procedure. During the study period, adverse events are collected through participants' symptom reports and researchers' observations, and the type of adverse event along with its causal relationship to the intervention is recorded in the Electronic Medical Record (EMR). In case of an adverse event, follow-up monitoring is conducted, and any severe adverse event is promptly reported. The causality of adverse events is classified into six levels based on the WHO-UMC causality categories: Certain (1), Probable/Likely (2), Possible (3), Unlikely (4), Conditional/Unclassified (5), and Unassessable/Unclassifiable (6).

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No